CLINICAL TRIAL: NCT00153673
Title: Phase III Study of a Double-Blind Randomized Comparison of Famotidine Plus Celecoxib Versus Dologesics for Gastric Ulcer Healing in Arthritis Patients (NSAID#5A Study)
Brief Title: Effect of Selective COX-2 Inhibition on Ulcer Healing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5NA study
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Arthritis; Gastric Ulcer
Keywords: celecoxib; arthritis; ulcer healing
MeSH Terms: conditions — Arthritis; Stomach Ulcer | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Celecoxib + Famotidine
  Interventions: Drug: celecoxib
- 2 (Active Comparator): Dologesics + Famotidine
  Interventions: Drug: Dologesics

INTERVENTIONS:
Drug: celecoxib — Celecoxib 200mg bd
  Arms: 1
Drug: Dologesics — Dologesics 2 tablets bd
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effect of Famotidine plus a COX-2 inhibitor (celecoxib) with Famotidine plus dologesics in ulcer healing in arthritis patients.

DETAILED DESCRIPTION:
For many years the integrity of the stomach mucosal barrier is thought to be maintained by mucosal prostaglandins (PG) synthesized by COX-1. However, the notion that COX-1 protects the stomach and COX-2 induces inflammation may be over-simplistic. In animal studies, COX-2, but not COX-1, is expressed in experimental gastric ulcer. Inhibition of COX-2 delays ulcer healing, indicating that PG derived from COX-2 contributes to restoring the mucosal barrier [1]. Whether this animal observation can be generalized to the human stomach is unknown. To date the biological functions of COX-1 and COX-2 in the healing of human gastric ulcer healing is unclear. Unlike experimental ulcers that only express COX-2, recently we have shown that both COX-1 and COX-2 are up-regulated in human gastric ulcers [2]. Furthermore, our preliminary results suggest that inhibition of COX-2 alone may not lead to a clinically significant delay in ulcer healing (refer to progress report). These observations suggest that peptic ulcer healing is more complex in the human stomach - both COX isoforms may be involved in the healing process. Inhibition of COX-2 alone may have less adverse effect than non-selective inhibition of both COX isoforms in ulcer healing. The current study aims to resolve the functional significance of COX-2 in human gastric ulcer from a biological and clinical perspective.

ELIGIBILITY:
Inclusion Criteria:

* Gastric ulcers confirmed by endoscopy
* Stop taking NSAIDs for 1 week prior to endoscopy
* Age 18
* H. pylori negative
* Informed written consent

Exclusion Criteria:

* Actively bleeding ulcers
* Ulcers showing dysplasia or malignancy
* Renal failure (serum creatinine >200umol/l)
* Previous gastric surgery
* Moribund or terminal malignancy
* Concomitant use of proton pump inhibitor, misoprostol, aspirin, steroid or anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2001-02; Primary Completion 2016-12-28 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
ulcer healing | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francis K Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, China